CLINICAL TRIAL: NCT00072982
Title: Treatment of Rheumatoid Arthritis With Marine and Botanical Oils
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Robert B. Zurier, MD, University of Massachusetts Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AT000309-01A2 (NIH); NIH RO1 AT000309-01A2; UMASS IRB Docket #10225; NEIRB Docket #04-039; FDA IND #69,292
Record Dates: First submitted 2003-11-13; First posted 2003-11-17 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Fish oil; Borage oil
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Fish Oils; borage oil; gamma-carboxyglutamyl-gamma-carboxyglutamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Fish Oil
  Interventions: Drug: fish oil
- 2 (Active Comparator): Borage Oil
  Interventions: Drug: borage seed oil
- 3 (Active Comparator): Fish Oil and Borage Oil
  Interventions: Drug: combination fish oil and borage seed oil

INTERVENTIONS:
Drug: fish oil — The object of this intervention is to determine whether treatment of rheumatoid arthritis with a combination of fish oil and borage seed oil is superior to treatment with either oil alone. Each arm of the study will take 13 capsules daily (divided doses) for 18 months.
  Other Names: EPA
  Arms: 1
Drug: borage seed oil — Borage oil 13 capsules divided doses daily for 18 months
  Other Names: GLA
  Arms: 2
Drug: combination fish oil and borage seed oil — Fish oil and borage seed oil capsules - 13 capsules to be be taken daily (divided doses) for a period of 18 months
  Other Names: EPA and GLA
  Arms: 3

SUMMARY:
The object of this study is to determine whether treatment of rheumatoid arthritis (RA) with a combination of fish oil and borage seed oil is superior to treatment with either oil alone. This study will also investigate the biochemical, immunological, and molecular mechanism responsible for the therapeutic effects of these fatty acids. Each patient will be followed for eighteen months.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria

* Definite RA with onset at > 16 years, with total disease duration of at least 6 months
* Active disease as manifested by at least 3 joints that are swollen and 6 joints that are tender at time of enrollment, and either an erythrocyte sedimentation rate >_28, or a CRP >1.4, or morning stiffness of at least 45 min
* Stable dose of DMARDs for 2 mos before baseline visit, with total duration of DMARD for 6 mos.
* All standard therapy for RA, including DMARDs and combinations of DMARDs will be allowed as long as doses have been stable for 2 mos
* Stable NSAID for 1 month before baseline if on an NSAID
* Stable prednisone dose of < 10 mg/day for 1 month before baseline visit, if on prednisone
* Ability to give and understand all elements of informed consent
* Absence of comorbid condition which, in the opinion of the physician-investigator, would render the patient unsuitable for the study
* Willingness to adhere to the clinical protocol.

Exclusion Criteria

* A diagnosis of inflammatory arthritis other than rheumatoid arthritis
* Chronic anticoagulation
* Hypersensitivity to fish or fish products or plant products
* A dose of prednisone of > 10 mg/day, or either a change in the prednisone dose or intra-articular corticosteroid injection within one month of the baseline evaluation
* An inability or unwillingness to use an effective form of contraception (females) during the duration of the study
* Pregnant and breast-feeding females
* Inability or unwillingness to adhere to the study diet
* Platelet count < 100,000/mm 3
* Hemoglobin < 9 g/dl
* Albumin < 3.3 g

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
The modified Disease Activity Score (DAS28) will be the primary outcome measure. | Assessed every 3 months

SECONDARY OUTCOMES:
Reduction of other medication for RA | Assessed every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Zurier, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (13):
- United States (13):
  - UAB Arthritis Clinical Intervention Program, Birmingham, Alabama
  - New England Res. Associates, Trumbull, Connecticut
  - RASF Clinical Research Center, Boca Raton, Florida
  - Lake Rheumatology, Tavares, Florida
  - Fallon Clinic Health Care, Worcester, Massachusetts
  - Division of Rheumatology, Umass Memorial Health Care, Worcester, Massachusetts
  - Rheumatology and Internal Medicine Associates of West County, PC, St Louis, Missouri
  - Joel M. Kremer, Albany, New York
  - Prem Tambar, MD, Niagara Falls, New York
  - Bryn Mawr Medical Specialists, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Piedmont Arthritis Clinic, Greenville, South Carolina